## **Statistical analysis Plan**

# TITLE: Process evaluation of the effectiveness of two transdiagnostic interventions targeting emotional regulation: compassion focused program and emotional skills training program

| N°ID RCB | N°CPP | N°CNIL |
|----------------|-----------------|---------|
| 2020-A00551-38 | 2020.09.03 ter_ | 2217007 |
| | 20.05.13.42837 | |

Document date: 17/01/2021

Study sponsor and investigator: Mathias Butaud, Psychiatrist 4 avenue Jean Perrot, 38000 Grenoble

**Co-investigator** : **Céline Baeyens**, Professor, Laboratoire Inter-universitaire de Psychologie, Université Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9

Associated investigators: Rebecca Bègue-Shankland, Professor au Laboratoire Développement, Individu, Processus, Handicap, Education (DIPHE), Université Lyon 2, Bâtiment V (V211 à V216), 5, Avenue Pierre Mendès-France, 69676 Bron Cedex, Marine Paucsik, PhD STudent, Laboratoire Interuniversitaire de Psychologie, Université Grenoble Alpes, UFR SHS, 1251 avenue Centrale, CS 40700, 38058 Grenoble Cedex 9, Francis Gheysen, psychiatrist, 1 avenue du 6 juin, 14000 Caen, Benjamin Gouache, psychiatrist, Claire Cécile Périer et Rocio Roure, neuropsychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble, Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères, Laure Favre-Réguillon, Psychologist – Centre Référent de Réhabilitation Psychosociale et de Remédiation cognitive (C3R) de Grenoble, Centre Ambulatoire de Santé Mentale, 8 place du Conseil de la Résistance, 38100 Saint-Martin-d'Hères, Céline Roussel, psychiatrist et Sandrine Rebelle, neuropsychologist, Centre départemental de réhabilitation psychosociale des Glières 219, Chemin des bois des Fornets 74800 La Roche-sur-Foron.

#### SINGLE CASE DESIGN

- Descriptive statistics (Kazdin, 2010)
- Pared sample T-test
- Intervention Time series analysis (ITSA)
- Tau-U

#### PILOT STUDY CLINICAL POPULATION

- T-test or Wilcoxon
- ANOVA (inter/intra and contrast)
- Regression analysis

### RANDOMIZED CONTROL STUDY SUBCLINICAL POPULATION

- T-test or Wilcoxon
- ANOVA (inter/intra and contrast)
- Regression analysis